CLINICAL TRIAL: NCT04736953
Title: Sirolimus Treatment of Patients With Systemic Lupus Erythematosus
Brief Title: Sirolimus Treatment Of Patients With SLE
Acronym: STOPSLE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Andras Perl, Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Rapamycin
Record Dates: First submitted 2020-12-04; First posted 2021-02-03 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Sirolimus; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sirolimus (Active Comparator): Sirolimus 1 to 2 mg bid
  Interventions: Drug: Sirolimus
- Placebo (Placebo Comparator): Placebo 1 to 2 mg bid
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sirolimus — Sirolimus
  Other Names: rapamycin
  Arms: Sirolimus
Other: Placebo — Placebo
  Other Names: Dextrose
  Arms: Placebo

SUMMARY:
Phase II Double-blind, placebo-controlled, randomized treatment trial with two arms: one SIROLIMUS arm with 92 patients and one placebo arm with 92 patients. The safety and therapeutic efficacy of SIROLIMUS will be determined within a dosage range of 1 mg/day to 4 mg/day, which will be titrated to tolerance during an initial 3-month open label period, relative to placebo in SLE patients over 12 months followed by a 1-month washout. The proposed study design, known as an enriched enrollment randomized withdrawal (EERW), has major advantages that (1) only people who tolerate SIROLIMUS are randomized, potentially reducing the percentage of dropouts in the randomized phase and (2) it allows participants to use an individualized dosage of study medication, which mimics clinical practice in terms of how SIROLIMUS would be administered. Healthy subjects receive no drugs and serve as controls for in vitro studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18;
2. Male or female;
3. ≥ 4 ACR SLE classification criteria;
4. Positive ANA at a titer of ≥ 1/80;
5. Stable immunosuppressants (MMF ≤ 3 g/day, azathioprine ≤ 100 mg/day; methotrexate ≤ 15 mg/day) and/or antimalarials (hydroxychloroquine ≤ 400 mg/day) for 30 days prior to screening; stable oral corticosteroids for 2 weeks prior to screening; ≤ 20 mg/day prednisone or equivalent; stable belimumab for 90 days prior to screening;
6. BILAG 2004 index (3) level A disease activity in ≥ 1 organ/system except renal or central nervous system or (ii) BILAG 2004 index level B disease activity in ≥ 2 organs/systems if no level A disease activity is present and (iii) SLEDAI ≥ 6;
7. Enrollment is approved by adjudication committee.

Exclusion Criteria:

1. Acute SLE flare threatening vital organs;
2. Pregnant or lactating;
3. Female subjects who are planning to become pregnant during the study or within 3 months after last dosing or male subjects who are considering fathering a child within 3 months after last dosing;
4. Abnormal laboratory test results: hemoglobin ≤ 8 g/L (8 g/dL), platelet count ≤ 70 x 109/L (70,000 cells/mm³), white blood cell count ≤ 2.0 x 109/L (2,000 cells/mm³), neutrophils: ≤ 1.5 X 109/L, proteinuria > 3 g/day measured by 24 hour collection or spot urine protein to creatinine ratio of >3;
5. Glomerular filtration rate (GFR) < 50 mL/min/1.73 m², any other clinically significant abnormal screening laboratory results as evaluated by the Investigator;
6. Moderately serious or serious comorbidities (e.g., diabetes mellitus, congestive heart failure, chronic obstructive pulmonary disease, chronic renal insufficiency) that in investigator's opinion confers high risk for adverse events;
7. Patients receiving cyclophosphamide within 3 months;
8. Active chronic infections (e.g., HIV, hepatitis B virus, hepatitis C virus, mycobacteria); patients with oral steroid-dependent asthma;
9. Infections requiring intravenous antibiotics within a month or oral antibiotics within two weeks of screening;
10. Patients taking (unwilling or unable to stop) NAC or other antioxidants within 1 month of screening (which is considered sufficient time to revert GSH to pre-treatment levels;
11. Patients receiving rituximab within 12 months or other biologic therapy within five half lives;
12. Patients receiving mTOR inhibitors (rapamycin/sirolimus, everolimus);
13. Patients enrolled in other interventional trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic Benefit | 12 months
  Positive Response on SLE Responder Index (SRI)